CLINICAL TRIAL: NCT04542421
Title: Lung Ultrasound Implementation in the Management of Patients Hospitalized With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-0781
Record Dates: First submitted 2020-09-04; First posted 2020-09-09 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: COVID-19; lung ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Lung ultrasound Implementation arm (Experimental): Hospitalists undergo training to use lung ultrasound in their patients hospitalized with COVID
  Interventions: Diagnostic Test: Lung ultrasound use in patients hospitalized with COVID

INTERVENTIONS:
Diagnostic Test: Lung ultrasound use in patients hospitalized with COVID — Hospitalists will be taught to use lung ultrasound in the management of their patients with COVID

SUMMARY:
Lung ultrasound (LUS) has also been shown to be more accurate than chest x-ray in identifying pulmonary consolidation and pulmonary edema, both of which are found in patients with COVID.

The investigators hypothesize implementation of LUS by hospitalists in the management of suspected or diagnosed patients with COVID-19 will reduce the need for Chest CT and chest x-ray, thereby conserving PPE, reducing risk of transmission to technicians and conserving the resources of radiology services that would otherwise be overwhelmed by patients with COVID-19 in need of chest imaging. Using the methods of implementation science, the investigators propose to respond to the urgent need for rapid implementation of LUS by hospitalists in management of adult patients hospitalized for COVID.

Aim 1a: Using a rapid-cycle weekly Plan-Do-Study-Act cycle and Rapid Iterative RE-AIM, to optimize the implementation of LUS by adult hospitalists in the management of COVID-19 patients in a pilot study

Aim 1b: Evaluate this pilot implementation of LUS by adult hospitalists using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

DETAILED DESCRIPTION:
Study overview:. The investigators will begin LUS implementation using strategies that target barriers already identified by hospitalists in prior qualitative work. The investigators will then proceed to conduct weekly rapid Plan-Do-Study-Act cycles informed by Rapid Iterative RE-AIM, in order to ensure timely identification of implementation barriers. Rapid Iterative RE- AIM is an innovative application of the RE-AIM framework in which screening assessments of RE-AIM outcomes (e.g. level of reach, adoption, implementation) which is performed at regular intervals during implementation and has been shown to be a feasible means of assessing interval implementation. For outcomes not meeting target implementation at our interval assessments, we will perform rapid qualitative interviews of key stakeholders to identify current barriers. Using the contextual domains of PRISM and rapid qualitative data from stakeholders we will select new or adapt existing implementation strategies, facilitating robust implementation. Study outcomes will be measured using the RE-AIM outcomes from PRISM including Reach, Effectiveness, Adoption, Implementation, and Maintenance.

Study Setting: University of Colorado Hospital is a 620 beds academic tertiary care center in Denver, Colorado.

Participant Recruitment: Hospitalist participants will be recruited from among the faculty of University of Colorado Hospital Division of hospital medicine which has over 100 physician and advanced practice clinicians (APPs).

Study Procedures:

All hospitalist physicians and APPs will be offered training in LUS. The training module to be used has been shown to be effective at training providers to competency. The investigators will evaluate acceptability and feasibility of the training module using rapid qualitative techniques and questionnaires of both completers and non-completers. Once a provider has completed training, she may begin performing LUS on COVID patients. The images will be wirelessly uploaded into PACS. The provider's LUS interpretation will be documented in the EMR. Rapid Iterative RE-AIM will be performed on a weekly basis as a means of iteratively screening for implementation barriers. The implementation outcomes of both fidelity and adaptation will be prioritized although all aspects of implementation will be evaluated. Interval Reach will be screened for using EMR data. For RE-AIM domains with poor implementation, the investigators will use rapid qualitative methods to obtain stakeholder perspectives of barriers and suggestions for adaptations to existing strategies or new strategies.

Measures/Data Collection Study Outcomes:

Reach: The investigators will measure the percentage of patients hospitalized with a positive COVID test result who received a LUS during the hospitalization. The investigators will compare the demographics and characteristics of the eligible patients who received a LUS versus those that did not in order to identify disparities in implementation that can be addressed by adapting our implementation strategies. The investigators will explore the underlying reasons for disparities in Reach using rapid qualitative interviews of providers and other stakeholders as appropriate.

Effectiveness: Using a quasi-experimental interrupted time series design, the investigators will compare the number of chest x-rays and CTs performed, PPE use and inpatient mortality in patient hospitalized with COVID before implementation of LUS versus after.

Adoption:

Adoption by clinicians will be measured by calculating the percentage of clinicians who completed the LUS training module within the UCH hospitalist group. The investigators will also measure the percentage of clinicians who performed at least 1 LUS exam. The investigators will evaluate for differences between providers who did and did not complete training. The investigators will interview hospitalists who did not complete training or did not perform LUS to understand why LUS was not adopted.

Implementation:

The investigators will focus on collecting implementation outcomes that are particularly relevant to the evaluation of diagnostic tests. Fidelity will be measured using data available through the EMR and through qualitative interviews of providers regarding their clinical decision-making. EMR data will be gathered by random selection of at least 10% of LUS exams within the EMR over the prior 30 days using the following 3 components to evaluate fidelity. 1. Image quality: Through the EMR, the investigators will assess whether image acquisition was adequate using a checklist of image requirements. 2. Image interpretation: the investigators will review interpretation of POCUS by assessing ultrasound reports in the EMR using a checklist 3. Clinical Decision-making using the LUS result: Assess appropriate integration of POCUS findings into the clinical decision-making by review of the LUS report in the EMR and daily clinician progress notes well as through qualitative interviews of providers.

Feasibility/Acceptability:

The investigators will measure feasibility and acceptability of the 1) LUS training module 2) use of LUS for evaluation of patients with COVID using a questionnaire as well as rapid qualitative interviews of hospitalists and other stakeholders

ELIGIBILITY:
Inclusion Criteria:

* Physicians and advanced care provider faculty in the Division of hospital medicine at University of Colorado Hospital, Aurora Colorado

Exclusion Criteria:

* Physicians and advanced care provider Faulty within the Division of Hospital medicine at University of Colorado Hospital who care for hospitalized patients less than 2 weeks per year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maw, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospitalists: 86 Hospitalists offered training to use lung ultrasound in their patients hospitalized with COVID. 4 out of 86 eligible hospitalists completed training and credentialing in lung ultrasound but all were followed throughout the 1 year study period
- Patients Hospitalized for COVID: 298 patients cared for by hospitalists received a lung ultrasound during 1 year period of data collection.
Period: Overall Study
Arm/Group | Hospitalists | Patients Hospitalized for COVID
Started | 86 | 298
Completed | 86 | 298
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Both Hospitalist and patients hospitalized for COVID were enrolled in this study
Groups:
- Hospitalists: All Hospitalists offered training to use lung ultrasound in their patients hospitalized with COVID 4 out of 86 eligible completed training and credentialing in lung ultrasound during 1 year period of data collection
- Patients Hospitalized for COVID: 298 patients hospitalized with COVID and cared for by a hospitalist
- Total: Total of all reporting groups
Arm/Group | Hospitalists | Patients Hospitalized for COVID | Total
Number analyzed (Participants) | 86 | 298 | 384
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 208 | 294
  >=65 years | 0 | 90 | 90
Age, Continuous [Mean (Full Range); unit: years] | 44 [31 to 54] | 57 [19 to 92] | 53 [19 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 134 | 183
  Male | 37 | 164 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 0 | 11 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 34 | 34
  White | 0 | 152 | 152
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 86 | 95 | 181
Region of Enrollment [Number; unit: participants]
  United States | 86 | 298 | 384
English speaking [Count of Participants; unit: Participants] | 86 | 214 | 300

OUTCOME MEASURES:

1. Primary Outcome: Hospitalists Who Adopt Lung Ultrasound
Description: Number of hospitalists who adopt lung ultrasound in the care of patients hospitalized with COVID
Time Frame: number of hospitalists who adopt lung ultrasound over a twelve month period
Measure: Count of Participants; unit: Participants
Groups:
- Lung Ultrasound Implementation Arm: hospitalists that adopt lung ultrasound over a 1 year period
Arm/Group | Lung Ultrasound Implementation Arm
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Patients With COVID Who Receive Lung Ultrasound
Description: patients with COVID who receive a lung ultrasound
Time Frame: patients with COVID who received a lung ultrasound by a hospitalist over a 12 month period
Measure: Count of Participants; unit: Participants
Groups:
- Lung Ultrasound Implementation Arm: All Hospitalists offered training to use lung ultrasound in their patients hospitalized with COVID. 4 out of 86 eligible hospitalists completed training and credentialing in lung ultrasound and 298 patients cared for by hospitalists received a lung ultrasound during 1 year period of data collection.
Arm/Group | Lung Ultrasound Implementation Arm
Number analyzed (Participants) | 298
Participants | 298

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Hospitalists Who Care for Patients With COVID: Hospitalists undergo training to use lung ultrasound in their patients hospitalized with COVID
- Patient Hospitalized With COVID: Patients hospitalized with COVID cared for by a hospitalist who received a lung ultrasound
Arm/Group | Hospitalists Who Care for Patients With COVID | Patient Hospitalized With COVID
All-Cause Mortality (participants affected / at risk) | 0/86 | 3/298
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/298
Other Adverse Events (participants affected / at risk) | 0/86 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04542421/Prot_SAP_000.pdf